CLINICAL TRIAL: NCT05573360
Title: Evaluation of Safety and Tolerability of Ocular Lubricants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DEE253-E001
Record Dates: First submitted 2022-10-04; First posted 2022-10-10 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sequence 1 (Other): NGF5-A/NGF4-B/NGF6-B/NGF6-E/Systane, 1 drop instilled to each eye, with a wash-out period of 1 to 7 days between each instillation
  Interventions: Other: NGF5-A test formulation; Other: NGF4-B test formulation; Other: NGF6-B test formulation; Other: NGF6-E test formulation; Other: Systane eye drop
- Sequence 2 (Other): NGF4-B/NGF6-B/NGF6-E/Systane/NGF5-A, 1 drop instilled to each eye, with a wash-out period of 1 to 7 days between each instillation
  Interventions: Other: NGF5-A test formulation; Other: NGF4-B test formulation; Other: NGF6-B test formulation; Other: NGF6-E test formulation; Other: Systane eye drop
- Sequence 3 (Other): NGF6-B/NGF6-E/Systane/NGF5-A/NGF4-B, 1 drop instilled to each eye, with a wash-out period of 1 to 7 days between each instillation
  Interventions: Other: NGF5-A test formulation; Other: NGF4-B test formulation; Other: NGF6-B test formulation; Other: NGF6-E test formulation; Other: Systane eye drop
- Sequence 4 (Other): NGF6-E/Systane/NGF5-A/NGF4-B/NGF6-B, 1 drop instilled to each eye, with a wash-out period of 1 to 7 days between each instillation
  Interventions: Other: NGF5-A test formulation; Other: NGF4-B test formulation; Other: NGF6-B test formulation; Other: NGF6-E test formulation; Other: Systane eye drop
- Sequence 5 (Other): Systane/NGF5-A/NGF4-B/NGF6-B/NGF6-E, 1 drop instilled to each eye, with a wash-out period of 1 to 7 days between each instillation
  Interventions: Other: NGF5-A test formulation; Other: NGF4-B test formulation; Other: NGF6-B test formulation; Other: NGF6-E test formulation; Other: Systane eye drop

INTERVENTIONS:
Other: NGF5-A test formulation — One drop of investigational product instilled on the eye
Other: NGF4-B test formulation — One drop of investigational product instilled on the eye
Other: NGF6-B test formulation — One drop of investigational product instilled on the eye
Other: NGF6-E test formulation — One drop of investigational product instilled on the eye
Other: Systane eye drop — One drop of commercial product instilled on the eye

SUMMARY:
The purpose of this study is to evaluate the safety profile of test formulations for an artificial tear product versus a comparator product.

DETAILED DESCRIPTION:
Subjects will be randomized to one of five different treatment sequences. Subjects will attend 6 scheduled visits with an expected individual duration of participation of 11 to 42 days. This study will be conducted in Australia.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an informed consent form.
* Willing and able to attend all study visits as required by the protocol.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any known active ocular disease.
* Any systemic condition that, in the opinion of the investigator, may affect a study outcome variable.
* Any ocular injury to either eye in the past 12 weeks prior to screening.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-Emergent Adverse Events (AEs) | Up to Day 30 (Study Exit)
  An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). The number of adverse events as observed or reported will be recorded.
Number of Subjects with Biomicroscopy Findings Outside of Normal Limits | Screening, up to Day 30 (Study Exit)
  The cornea, conjunctiva, and eyelid will be assessed using a slit lamp. The number of subjects with biomicroscopy findings outside of normal limits will be recorded.
Mean Total Ocular Surface Staining Score | Screening, up to Day 30 (Study Exit)
  Ocular surface staining will be assessed using a slit lamp and recorded on a 15-point scale.
Mean Best Corrected Visual Acuity (BCVA) | Screening, up to Day 30 (Study Exit)
  Visual Acuity will be assessed with correction in place using letter charts. BCVA will be measured in logarithm Minimum Angle of Resolution (logMAR).
Number of Device Deficiencies | Up to Day 30 (Study Exit)
  A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. The number of device deficiencies as observed or reported will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Dry Eye, Study Director — Alcon Research, LLC
Locations (2):
- Australia (2):
  - Alcon Investigator 8169, Carlton, Victoria
  - Alcon Investigator 8214, Waurn Ponds, Victoria

IPD SHARING:
Plan to Share IPD: No